CLINICAL TRIAL: NCT03952039
Title: A Phase 3, Multicenter, Open-label, Randomized Study to Evaluate the Efficacy and Safety of Fedratinib Compared to Best Available Therapy (BAT) in Subjects With DIPSS (Dynamic International Prognostic Scoring System)-Intermediate or High-risk Primary Myelofibrosis (PMF), Post-polycythemia Vera Myelofibrosis (Post-PV MF), or Post-essential Thrombocythemia Myelofibrosis (Post-ET MF) and Previously Treated With Ruxolitinib
Brief Title: An Efficacy and Safety Study of Fedratinib Compared to Best Available Therapy in Subjects With DIPSS-intermediate or High-risk Primary Myelofibrosis, Post-polycythemia Vera Myelofibrosis, or Post-essential Thrombocythemia Myelofibrosis and Previously Treated With Ruxolitinib
Acronym: FREEDOM2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Impact Biomedicines, Inc., a wholly owned subsidiary of Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEDR-MF-002; U1111-1223-2962 (Registry Identifier: WHO); 2018-003411-21 (EudraCT Number)
Expanded Access: NCT03723148 (Available)
Record Dates: First submitted 2019-05-06; First posted 2019-05-16 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera; Myelofibrosis
Keywords: MF; myeloproliferative neoplasms; MPN; myelofibrosis; PMF; post-PV; Post-Polycythemia Vera; post-ET MF; Post-Essential Thrombocythemia Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fedratinib 400mg/day (Experimental): Will include up to 128 subjects receiving fedratinib 400 mg self-administered Investigational Product (IP) on an outpatient basis, once daily preferably together with food during an evening meal at the same time each day in consecutive 4-week (28-day) cycles.
  Interventions: Drug: FEDRATINIB
- Best Available Therapy (BAT) (Active Comparator): Best-available Investigator-selected therapy included a number of available compounds to treat MF and/or its symptoms and was chosen by the investigator for each subject. Therapy changed at different times during the treatment period. No investigational agents (e.g. not approved for the treatment of any indication) were allowed. BAT also included the choice of no treatment.
  Interventions: Drug: Best Available Therapy (BAT)

INTERVENTIONS:
Drug: FEDRATINIB — A potent and selective inhibitor of JAK2 kinase activity
  Arms: Fedratinib 400mg/day
Drug: Best Available Therapy (BAT) — Best available therapy (BAT)
  Arms: Best Available Therapy (BAT)

SUMMARY:
A Phase 3, multicenter, open-label, randomized study to evaluate the efficacy and safety of fedratinib compared to best available therapy (BAT) in subjects with DIPSS (Dynamic International Prognostic Scoring System)-intermediate or high-risk primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (post-PV MF), or post-essential thrombocythemia myelofibrosis (post-ET MF) and previously treated with ruxolitinib. The primary objective of the study is to evaluate the percentage of subjects with at least 35% spleen volume reduction in the fedratinib and the BAT arms.

DETAILED DESCRIPTION:
This Phase 3, multicenter, randomized, two-arm, open-label study will include subjects with intermediate or high-risk (as per the DIPSS score) primary myelofibrosis (PMF), postpolycythemia vera myelofibrosis (post-PV MF), or post-essential thrombocythemia myelofibrosis (post-ET MF). This study will be conducted in compliance with International Council for Harmonisation (ICH) Good Clinical Practices (GCPs).

Study design includes:

* A 28-day Screening Period
* 2:1 Randomization to fedratinib or best available therapy (BAT)
* Stratification at Randomization according to:

  * Spleen size by palpation: < 15 cm below left costal margin (LCM) versus ≥ 15 cm below LCM
  * Platelets ≥ 50 to < 100 x 109/L versus platelets ≥ 100 x 109/L
  * Refractory or relapsed to ruxolitinib treatment versus intolerant to ruxolitinib treatment
* Study Treatment Period (time on study drug plus 30 days after last dose)
* Subjects are allowed to crossover from BAT to the fedratinib arm after the Cycle 6 response assessment or before the Cycle 6 response assessment in the event of a confirmed progression of splenomegaly by MRI/CT scan
* A Survival Follow-up Period for progression and survival

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age at the time of signing the informed consent form (ICF)
2. Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) of 0, 1 or 2
3. Subject has diagnosis of primary myelofibrosis (PMF) according to the 2016 World Health Organization (WHO) criteria, or diagnosis of post-ET or post-PV myelofibrosis according to the IWG-MRT 2007 criteria, confirmed by the most recent local pathology report
4. Subject has a DIPSS Risk score of Intermediate-2 or High
5. Subject has a measurable splenomegaly during the screening period as demonstrated by spleen volume of ≥ 450 cm3 by MRI or CT-scan and by palpable spleen measuring ≥ 5 cm below the left costal margin
6. Subject has a measurable total symptoms score (≥ 1) as measured by the Myelofibrosis Symptom Assessment Form (MFSAF)
7. Subject has been previously exposed to ruxolitinib, and must meet at least one of the following criteria (a and/or b)

   1. Treatment with ruxolitinib for ≥ 3 months with inadequate efficacy response (refractory) defined as < 10% spleen volume reduction by MRI or < 30% decrease from baseline in spleen size by palpation or regrowth (relapsed) to these parameters following an initial response
   2. Treatment with ruxolitinib for ≥ 28 days complicated by any of the following (intolerant):

      * Development of a red blood cell transfusion requirement (at least 2 units/month for 2 months) or
      * Grade ≥ 3 AEs of thrombocytopenia, anemia, hematoma, and/or hemorrhage while on treatment with ruxolitinib
8. Subject must have treatment-related toxicities from prior therapy resolved to Grade 1 or pretreatment baseline before start of last therapy prior to randomization
9. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted
10. Subject is willing and able to adhere to the study visit schedule and other protocol requirements
11. A female of childbearing potential (FCBP) must:

    1. Have 2 negative pregnancy tests as verified by the Investigator during screening prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
    2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use and be able to comply with highly effective contraception without interruption, -14 days prior to starting investigational product, during the study treatment (including dose interruptions), and for 30 days after discontinuation of study treatment.

    Note: A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
12. A male subject must:

Practice true abstinence (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 30 days following investigational product discontinuation, or longer if required for each compound and/or by local regulations, even if he has undergone a successful vasectomy

Exclusion Criteria:

1. Any of the following laboratory abnormalities:

   1. Platelets < 50 x 109/L
   2. Absolute neutrophil count (ANC) < 1.0 x 109/L
   3. White blood count (WBC) > 100 x 109/L
   4. Myeloblasts ≥ 5 % in peripheral blood
   5. Estimated glomerular filtration rate < 30 mL/min/1.73 m2 (as per the Modification of Diet in Renal Disease [MDRD] formula)
   6. Serum amylase or lipase > 1.5 x upper limit of normal (ULN)
   7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN)
   8. Total bilirubin > 1.5 x ULN, subject's total bilirubin between 1.5 - 3.0 x ULN are eligible if the direct bilirubin fraction is < 25% of the total bilirubin
2. Subject is pregnant or lactating female
3. Subject with previous splenectomy
4. Subject with previous or planned hematopoietic cell transplant
5. Subject with prior history of encephalopathy, including Wernicke's (WE)
6. Subject with signs or symptoms of encephalopathy, including WE (eg, severe ataxia, ocular paralysis or cerebellar signs)
7. Subject with thiamine deficiency, defined as thiamine levels in whole blood below normal range according to the central laboratory and not demonstrated to be corrected prior to randomization
8. Subject with concomitant treatment with or use of pharmaceutical, herbal agents or food known to be strong or moderate inducers of Cytochrome P450 3A4 (CYP3A4), or dual CYP2C19 and CYP3A4 inhibitors
9. Subject on any chemotherapy, immunomodulatory drug therapy (eg, thalidomide, interferon-alpha), anagrelide, immunosuppressive therapy, systemic corticosteroids > 10 mg/day prednisone or equivalent. Subjects who have had prior exposure to hydroxyurea (eg, Hydrea) in the past may be enrolled into the study as long as it has not been administered within 14 days prior to randomization
10. Subject has received ruxolitinib within 14 days prior to randomization
11. Subject with previous exposure to Janus kinase (JAK) inhibitor(s) other than ruxolitinib treatment
12. Subject on treatment with aspirin with doses > 150 mg daily
13. Subject with major surgery within 28 days prior to randomization
14. Subject with diagnosis of chronic liver disease (eg, chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemochromatosis, non-alcoholic steatohepatitis)
15. Subject with prior malignancy other than the disease under study unless the subject has not required treatment for the malignancy for at least 3 years prior to randomization. However, subject with the following history/concurrent conditions provided successfully treated may enroll: non-invasive skin cancer, in situ cervical cancer, carcinoma in situ of the breast, incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system), or is free of disease and on hormonal treatment only
16. Subject with uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4)
17. Subject with known human immunodeficiency virus (HIV), known active infectious Hepatitis B (HepB), and/or known active infectious Hepatitis C (HepC)
18. Subject with serious active infection
19. Subject with presence of any significant gastric or other disorder that would inhibit absorption of oral medication
20. Subject is unable to swallow capsule
21. Subject with any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
22. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
23. Subject has any condition that confounds the ability to interpret data from the study
24. Subject with participation in any study of an investigational agent (drug, biologic, device) within 30 days prior to randomization
25. Subject with a life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2025-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (107):
- Australia (5):
  - Local Institution - 103, Darlinghurst, New South Wales
  - Local Institution - 101, Adelaide, South Australia
  - Local Institution - 105, Box Hill, Victoria
  - Local Institution - 102, Langwarrin, Victoria
  - Local Institution - 100, Melbourne
- Austria (7):
  - Local Institution - 156, Graz
  - Local Institution - 154, Innsbruck
  - Local Institution - 155, Linz
  - Local Institution - 151, Salzburg
  - Local Institution - 150, Vienna
  - Local Institution - 152, Vienna
  - Local Institution - 153, Wels
- Belgium (6):
  - Local Institution - 200, Bruges
  - Local Institution - 202, Brussels
  - Local Institution - 205, La Louvière-(Haine St-Paul)
  - Local Institution - 201, Leuven
  - Local Institution - 204, Liège
  - Local Institution - 203, Yvoir
- China (4):
  - Local Institution - 555, Beijing
  - Local Institution - 550, Guangzhou, Guangdong
  - Local Institution - 553, Tianjin
  - Local Institution - 557, Zhengzhou
- Czechia (3):
  - Local Institution - 700, Brno
  - Local Institution - 702, Ostrava-Poruba
  - Local Institution - 701, Prague
- France (12):
  - Local Institution - 255, Angers
  - Local Institution - 256, Brest
  - Local Institution - 254, Lens
  - Local Institution - 259, Lille
  - Local Institution - 260, Nice
  - Local Institution - 250, Nîmes
  - Local Institution - 252, Paris
  - Local Institution - 258, Pessac
  - Local Institution - 257, Pierre-Bénite
  - Local Institution - 261, Poitiers
  - Local Institution - 251, Strasbourg
  - Local Institution - 253, Toulouse
- Germany (8):
  - Local Institution - 302, Aachen
  - Local Institution - 308, Frankfurt am Main
  - Local Institution - 306, Halle
  - Local Institution - 303, Jena
  - Local Institution - 307, Magdeburg
  - Local Institution - 301, Mannheim
  - Local Institution - 304, Minden
  - Local Institution - 305, Ulm
- Hungary (5):
  - Local Institution - 600, Budapest
  - Local Institution - 601, Győr
  - Local Institution - 602, Kaposvár
  - Local Institution - 604, Nyíregyháza
  - Local Institution - 603, Szeged
- Ireland (3):
  - Local Institution - 751, Cork
  - Local Institution - 752, Dublin
  - Local Institution - 750, Dublin
- Italy (14):
  - Local Institution - 353, Bologna
  - Local Institution - 363, Brescia
  - Local Institution - 354, Catania
  - Local Institution - 350, Florence
  - Local Institution - 358, Milan
  - Local Institution - 362, Naples
  - Local Institution - 357, Pavia
  - Local Institution - 356, Roma
  - Local Institution - 361, Roma
  - Local Institution - 359, Roma
  - Local Institution - 355, Torino
  - Local Institution - 360, Udine
  - Local Institution - 352, Varese
  - Local Institution - 364, Verona
- Netherlands (2):
  - Local Institution - 402, Maastricht
  - Local Institution - 400, Nijmegen
- Poland (3):
  - Local Institution - 803, Poznan
  - Local Institution - 801, Warsaw
  - Local Institution - 802, Wroclaw
- Russia (8):
  - Local Institution - 855, Moscow
  - Local Institution - 851, Moscow
  - Local Institution - 853, Moscow
  - Local Institution - 857, Novosibirsk
  - Local Institution - 852, Saint Petersburg
  - Local Institution - 854, Saint Petersburg
  - Local Institution - 850, Saint Petersburg
  - Local Institution - 859, Vladikavkaz
- South Korea (6):
  - Local Institution - 900, Seongnam-si
  - Local Institution - 905, Seoul
  - Local Institution - 901, Seoul
  - Local Institution - 903, Seoul
  - Local Institution - 904, Seoul
  - Local Institution - 902, Seoul
- Spain (14):
  - Local Institution - 451, Alicante
  - Local Institution - 452, Badalona (Barcelona)
  - Local Institution - 458, Barakaldo
  - Local Institution - 450, Barcelona
  - Local Institution - 462, Girona
  - Local Institution - 461, Las Palmas de Gran Canaria
  - Local Institution - 453, Madrid
  - Local Institution - 459, Madrid
  - Local Institution - 457, Málaga
  - Local Institution - 454, Murcia
  - Local Institution - 455, Salamanca
  - Local Institution - 463, Santa Cruz de Tenerife
  - Local Institution - 460, Santiago de Compostela
  - Local Institution - 456, Valencia
- United Kingdom (7):
  - Local Institution - 504, Manchester, Lancashire
  - Local Institution - 506, Nottingham, Nottinghamshire
  - Local Institution - 502, Birmingham
  - Local Institution - 503, Boston
  - Local Institution - 501, London
  - Local Institution - 505, London
  - Local Institution - 500, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Harrison CN, Mesa R, Talpaz M, Al-Ali HK, Xicoy B, Passamonti F, Palandri F, Benevolo G, Vannucchi AM, Mediavilla C, Iurlo A, Kim I, Rose S, Brown P, Hernandez C, Wang J, Kiladjian JJ. Efficacy and safety of fedratinib in patients with myelofibrosis previously treated with ruxolitinib (FREEDOM2): results from a multicentre, open-label, randomised, controlled, phase 3 trial. Lancet Haematol. 2024 Oct;11(10):e729-e740. doi: 10.1016/S2352-3026(24)00212-6. Epub 2024 Sep 9. PMID 39265613
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 201 participants randomized and treated
Groups:
- Fedratinib: Fedratinib 400mg/Day PO(4x100mg capsules)
- Best Available Therapy (BAT): Best available therapy regimen (BAT) may include any Investigator-selected treatment and is not limited to approved JAK inhibitors (used according to the prescribing information), chemotherapy (eg, hydroxyurea), anagrelide, corticosteroid, hematopoietic growth factor, immunomodulating agent, androgens, interferon, and may also include "no treatment" and symptom directed treatment. BAT may not include investigational agents, fedratinib (if approved during the course of the study) and hematopoietic stem cell transplantation.
Period: Overall Study
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Started | 134 | 67
Participants Who Crossed Over | 0 | 46
Completed (Completed = Treatment ongoing) | 43 | 28
Not Completed | 91 | 39
Not completed — Adverse Event | 22 | 8
Not completed — Withdrawal by Participant | 17 | 12
Not completed — Death | 13 | 6
Not completed — Lack of Efficacy | 12 | 2
Not completed — Physician Decision | 9 | 3
Not completed — Progressive Disease | 6 | 4
Not completed — Other Reasons | 12 | 4

BASELINE CHARACTERISTICS:
Population: Intent to Treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Fedratinib | Best Available Therapy (BAT) | Total
Number analyzed (Participants) | 134 | 67 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (8.79) | 67.6 (8.16) | 68.4 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 37 | 96
  Male | 75 | 30 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 106 | 57 | 163
  Unknown or Not Reported | 20 | 7 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 106 | 58 | 164
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Spleen Volume Response Rate (RR)
Description: Percentage of participants who have ≥ 35% spleen volume reduction (SVR) at end of cycle 6
  A Cochran-Mantel-Haenszel (CMH) test to adjust for planned stratification factors (spleen size by palpation, platelet counts and refractory/relapsed or intolerance to ruxolitinib treatment).
  The RRs and 95% confidence intervals (CI) will be provided for each arm as well as for the difference in RRs and 95% confidence interval of the difference for fedratinib to BAT.
Time Frame: From Screening to end of Cycle 6 (1 cycle = 28 days), approximately 196 days
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 134 | 67
Percentage of Participants | 35.8 [27.7 to 44.6] | 6.0 [1.7 to 14.6]
Statistical Analysis 1: Comparison: Fedratinib vs Best Available Therapy (BAT); Stratified analysis (based on CRF); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test using the Greenland and Robins method to adjust for stratification factors: spleen size by palpation and platelet counts; Difference in Proportion = 29.6, 95% CI 2-sided [19.9 to 39.4]

2. Secondary Outcome: Symptom Response Rate (SRR)
Description: Percentage of participants with ≥ 50% reduction in total symptom scores measured by Myelofibrosis Symptom Assessment Form (MFSAF) 4.0 at end of cycle 6.
  Subjects with a missing TSS at the end of cycle 6 or who had disease progression before the end of the cycle 6 will be considered non-responders.
  MFSAF measures the sum of 7 symptoms on a scale from 0 to 10 (0 being absent and 10 being the worst imagineable). The lower the score the better.
  A Cochran-Mantel-Haenszel (CMH) test to adjust for planned stratification factors (spleen size by palpation, platelet counts and refractory/relapsed or intolerance to ruxolitinib treatment).
  The SRRs and 95% confidence intervals (CI) will be provided for each arm as well as for the difference in SRRs and 95% confidence interval of the difference for fedratinib to BAT.
Time Frame: From Cycle 1 Dose 1 to end of Cycle 6, approximately 168 days
Population: ITT population with non-zero baseline TSS
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 126 | 65
Percentage of Participants | 34.1 [25.9 to 43.1] | 16.9 [8.8 to 28.3]
Statistical Analysis 1: Comparison: Fedratinib vs Best Available Therapy (BAT); Test type: Superiority — Stratified analysis (based on CRF); p = 0.0033, Cochran-Mantel-Haenszel; CMH test using the Greenland and Robins method to adjust for stratification factors: spleen size by palpation and platelet counts; Difference in Proportion = 17.1, 95% CI 2-sided [4.8 to 29.4]

3. Secondary Outcome: Spleen Volume Response Rate (RR25)
Description: Percentage of participants who have ≥ 25% spleen volume reduction (SVR) at end of cycle 6
  A Cochran-Mantel-Haenszel (CMH) test to adjust for planned stratification factors (spleen size by palpation, platelet counts and refractory/relapsed or intolerance to ruxolitinib treatment).
  The RRs and 95% confidence intervals (CI) will be provided for each arm as well as for the difference in RRs and 95% confidence interval of the difference for fedratinib to BAT.
Time Frame: From Screening to end of Cycle 6 (1 cycle = 28 days), approximately 196 days
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 134 | 67
Percentage of Participants | 47.0 [38.3 to 55.8] | 13.4 [6.3 to 24.0]
Statistical Analysis 1: Comparison: Fedratinib vs Best Available Therapy (BAT); Stratified analysis (based on CRF); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in Proportion = 33.5, 95% CI 2-sided [21.9 to 45.1]

4. Secondary Outcome: Number of Participants With All Grade Treatment Emergent Adverse Events (AEs) and Grade 3 to 4 Treatment Emergent AEs
Description: Number of participants with all grade adverse events (AEs) and grade 3 to 4 AEs
Time Frame: From Cycle 1 Dose 1 to end of Cycle 6, approximately 168 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 134 | 67
Participants
  All Grade AEs | 132 | 65
  Grade 3 and 4 AEs | 88 | 29

5. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities
Description: Number of participants with hematology laboratory abnormalities in the following parameters: hemoglobin (decreased), leukocytes (increase and decrease), lymphocytes (decreased), neutrophils (segmented and band form decreased), Platelets (decreased).
Time Frame: From Cycle 1 Dose 1 to end of Cycle 6, approximately 168 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 134 | 67
Participants
  Hemoglobin Decreased All Grades: number analyzed (Participants) | 131 | 65
  Hemoglobin Decreased All Grades | 129 | 64
  Hemoglobin Decreased Grade 3: number analyzed (Participants) | 131 | 65
  Hemoglobin Decreased Grade 3 | 62 | 20
  Hemoglobin Decreased Grade 4: number analyzed (Participants) | 131 | 65
  Hemoglobin Decreased Grade 4 | 0 | 0
  Leukocytes Decreased All Grades: number analyzed (Participants) | 131 | 65
  Leukocytes Decreased All Grades | 41 | 19
  Leukocytes Decreased Grade 3: number analyzed (Participants) | 131 | 65
  Leukocytes Decreased Grade 3 | 8 | 3
  Leukocytes Decreased Grade 4: number analyzed (Participants) | 131 | 65
  Leukocytes Decreased Grade 4 | 1 | 0
  Leukocytes Increased All Grades: number analyzed (Participants) | 131 | 65
  Leukocytes Increased All Grades | 4 | 4
  Leukocytes Increased Grade 3: number analyzed (Participants) | 131 | 65
  Leukocytes Increased Grade 3 | 4 | 4
  Leukocytes Increased Grade 4: number analyzed (Participants) | 131 | 65
  Leukocytes Increased Grade 4 | 0 | 0
  Lymphocytes Decreased All Grades: number analyzed (Participants) | 129 | 64
  Lymphocytes Decreased All Grades | 49 | 20
  Lymphocytes Decreased Grade 3: number analyzed (Participants) | 129 | 64
  Lymphocytes Decreased Grade 3 | 20 | 7
  Lymphocytes Decreased Grade 4: number analyzed (Participants) | 129 | 64
  Lymphocytes Decreased Grade 4 | 1 | 0
  Neutrophils, segmented and band from decreased All Grades: number analyzed (Participants) | 129 | 64
  Neutrophils, segmented and band from decreased All Grades | 34 | 15
  Neutrophils, segmented and band from decreased Grade 3: number analyzed (Participants) | 129 | 64
  Neutrophils, segmented and band from decreased Grade 3 | 11 | 4
  Neutrophils, segmented and band from decreased Grade 4: number analyzed (Participants) | 129 | 64
  Neutrophils, segmented and band from decreased Grade 4 | 0 | 0
  Platelets Decreased All Grades: number analyzed (Participants) | 125 | 62
  Platelets Decreased All Grades | 73 | 43
  Platelets Decreased Grade 3: number analyzed (Participants) | 125 | 62
  Platelets Decreased Grade 3 | 24 | 10
  Platelets Decreased Grade 4: number analyzed (Participants) | 125 | 62
  Platelets Decreased Grade 4 | 3 | 2

6. Secondary Outcome: Spleen Response Rate by Palpation (RRP)
Description: Spleen response rate by palpation is the percentage of participants at the end of cycle 6 with a spleen response according to the IWG-MRT 2013 criteria.
  A baseline splenomegaly that is palpable at 5-10 cm, below the LCM, becomes not palpable** or A baseline splenomegaly that is palpable at > 10 cm, below the LCM, decreases by ≥ 50%**
  Participants with a missing spleen size assessment at the end of cycle 6 including those who meet the criteria for progression of splenomegaly before end of cycle 6 will be considered not to be responders.
Time Frame: From Cycle 1 Dose 1 to end of Cycle 6, approximately 168 days
Population: Intent to Treat Population with baseline spleen size ≥5 cm below the lower costal margin (LCM)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 134 | 65
Percentage of Participants | 28.4 [20.9 to 36.8] | 7.7 [2.5 to 17.0]
Statistical Analysis 1: Comparison: Fedratinib vs Best Available Therapy (BAT); Test type: Superiority; Greenland and Robins method; Greenland and Robins method = 19.9, 95% CI 2-sided [10.0 to 29.7]

7. Secondary Outcome: Durability of Spleen Volume Response (DR)
Description: Durability of spleen volume response (DR) by MRI/CT is defined as the date from the first documented spleen response (ie, ≥ 35% reduction in spleen volume) to the date of subsequent progressive disease (PD) in spleen volume per the IWG-MRT 2013 criteria or death, whichever is earlier. In the absence of an event before the analysis is performed, the DR will be censored at the date of the last valid assessment performed before the analysis performed date.
Time Frame: From baseline to end of treatment visit, Approximately on average 53 weeks up to 151 weeks.
Population: Participants with spleen volume response at any time
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 72 | 8
Weeks | 86.3 [63.0 to 126.4] | NA [NA to NA] — Median, lower limit number and upper limit number are not estimable due to an insufficient number of events needed to calculate via KM methodology.

8. Secondary Outcome: Durability of Spleen Response by Palpation (DRP)
Description: Durability of spleen response by palpation (DRP) is defined as time from the date of the first documented palpable spleen response, according to the IWG-MRT 2013 to the date of the subsequent PD in spleen size according to the IWG-MRT 2013 or death, whichever is earlier. Durability of spleen response by palpation according to the IWG-MRT 2013 criteria will be calculated for subjects that have an enlarged spleen at baseline (≥ 5 cm below LCM), and that have a spleen response by palpation. In the absence of an event before the analysis is performed, the DRP will be censored at the date of the last valid assessment performed before the analysis performed date.
Time Frame: From baseline to end of treatment visit, Approximately on average 53 weeks up to 151 weeks.
Population: Participants with spleen response by palpation at any time
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 71 | 11
Weeks | 118.3 [76.0 to NA] — The upper limit number is not estimable due to an insufficient number of events needed to calculate via KM methodology. | 47.1 [21.7 to NA] — The upper limit number is not estimable due to an insufficient number of events needed to calculate via KM methodology.

9. Secondary Outcome: Durability of Symptoms Response (DSR)
Description: The DSR is defined as time from the first documented response in TSS (ie, reduction in TSS ≥ 50%) measured by MFSAF version 4.0 to the first documented TSS reduction < 50%. In the absence of TSS reduction < 50% before the analysis performed, the DSR will be censored at the date of the last valid assessment performed before the analysis performed date.
Time Frame: From baseline to end of treatment visit, Approximately on average 53 weeks up to 151 weeks.
Population: Participants with a symptom response at any time
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 90 | 32
Weeks | 12.1 [8.1 to 16.1] | 10.1 [4.1 to 16.7]

10. Secondary Outcome: Assessment of the Effectiveness of Risk Mitigation Strategy for ≥3 Grade Gastrointestinal Adverse Events and Any Grade Wernickes Encephalopathy
Description: Number of participants with a CTCAE Grade ≥3 of nausea, diarrhea, or vomiting and any grade wernickes encephalopathy.
Time Frame: From Screening to end of Cycle 6 (1 cycle = 28 days), approximately 196 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 134 | 67
Participants
  ≥3 grade Diarrhea | 2 | 0
  ≥3 grade Nausea | 1 | 0
  ≥3 grade Vomitting | 0 | 0
  Any Grade Wernickes Encephalopathy | 1 | 0

11. Secondary Outcome: Number of Participants With Thiamine Levels Below the Lower Limit of Normal
Description: Number of participants with thiamine levels below the lower limit of normal
Time Frame: From Cycle 1 Dose 1 to end of Cycle 6, approximately 168 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 134 | 67
Participants
  Cycle 1 | 3 | 0
  Cycle 2: number analyzed (Participants) | 121 | 58
  Cycle 2 | 13 | 0
  Cycle 3: number analyzed (Participants) | 117 | 58
  Cycle 3 | 11 | 1
  Cycle 4: number analyzed (Participants) | 71 | 26
  Cycle 4 | 1 | 0
  Cycle 5: number analyzed (Participants) | 45 | 15
  Cycle 5 | 1 | 0
  Cycle 6: number analyzed (Participants) | 97 | 55
  Cycle 6 | 2 | 1

12. Secondary Outcome: Mean Change in EORTC QOL-C30 at Cycle 7 Day 1 as Compared With Baseline
Description: QLQ-C30 - The EORTC QLQ-C30 was developed to assess the quality of life of cancer patients. It consists of 30 items classified into 15 domains including 5 functional subscales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning); 3 multi-item symptom subscales (fatigue, nausea/vomiting, and pain); a global QOL subscale; and 6 single items addressing various symptoms and perceived financial impact. Scores vary from 0 (worst) to 100 (best) for the functional dimensions and GHS, and from 0 (best) to 100 (worst) for the symptom dimensions.
Time Frame: from the start of cycle 1 to cycle 7 day 1 approximately 170 days.
Population: EORTC QOL-C30 evaluable population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 105 | 50
Scores on a Scale
  Global Heath Status: number analyzed (Participants) | 69 | 21
  Global Heath Status | 10.3 (27.42) | 13.1 (26.16)
  Physical Functioning: number analyzed (Participants) | 70 | 21
  Physical Functioning | 8.2 (19.57) | 11.1 (26.61)
  Role Functioning: number analyzed (Participants) | 70 | 21
  Role Functioning | 8.1 (34.26) | 12.7 (40.79)
  Emotional Functioning: number analyzed (Participants) | 69 | 21
  Emotional Functioning | 7.0 (19.63) | 5.6 (25.86)
  Cognitivie Functioning: number analyzed (Participants) | 69 | 21
  Cognitivie Functioning | 1.7 (19.83) | 5.6 (17.74)
  Social Functioning: number analyzed (Participants) | 69 | 21
  Social Functioning | 6.5 (29.18) | 0.0 (27.89)
  Fatigue: number analyzed (Participants) | 70 | 21
  Fatigue | -15.2 (29.34) | -16.4 (33.81)
  Nausea and Vomitting: number analyzed (Participants) | 70 | 21
  Nausea and Vomitting | -1.7 (15.32) | -9.5 (28.17)
  Pain: number analyzed (Participants) | 70 | 21
  Pain | -12.9 (25.88) | -9.5 (33.57)
  Dyspnea: number analyzed (Participants) | 70 | 21
  Dyspnea | -9.0 (31.04) | -22.2 (35.49)
  Insomnia: number analyzed (Participants) | 70 | 21
  Insomnia | -11.4 (30.50) | -7.9 (25.61)
  Appetite Loss: number analyzed (Participants) | 70 | 21
  Appetite Loss | -19.5 (32.84) | -20.6 (35.71)
  Constipation: number analyzed (Participants) | 70 | 21
  Constipation | -0.5 (31.34) | -9.5 (35.19)
  Diarrhea: number analyzed (Participants) | 69 | 21
  Diarrhea | 5.3 (27.19) | 6.3 (17.06)
  Financial Difficulties: number analyzed (Participants) | 69 | 21
  Financial Difficulties | 3.9 (21.03) | 1.6 (12.81)

13. Secondary Outcome: Mean Change From Baseline in EQ-5D-5L Utility Index Score
Description: EQ-5D-5L - The EQ-5D-5L is a generic, self-administered preference-based measure of health. The five dimensions covered by the EQ-5D-5L include mobility, self-care, pain, usual activities, and anxiety/depression and is converted into a single summary index that can range from -0.594 to 1.0, with a score of 0 indicating death, 1.00 indicating "full health," and negative scores reflecting states perceived to be worse than death. Respondent's self-rated health on a vertical, 0 to 100 scale where 100 = "Best imaginable health state" and 0 = "Worst imaginable health state"
Time Frame: from the start of cycle 1 to cycle 7 day 1 approximately 170 days.
Population: EQ-5D-5L evaluable population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Fedratinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 103 | 52
Scores on a Scale
  C2D1: number analyzed (Participants) | 94 | 41
  C2D1 | 0.1086 (0.20188) | 0.0705 (0.22881)
  C3D1: number analyzed (Participants) | 88 | 48
  C3D1 | 0.1093 (0.23950) | 0.1142 (0.26247)
  C4D1: number analyzed (Participants) | 84 | 43
  C4D1 | 0.1214 (0.20634) | 0.0366 (0.26470)
  C5D1: number analyzed (Participants) | 78 | 43
  C5D1 | 0.1068 (0.21395) | 0.0321 (0.23607)
  C6D1: number analyzed (Participants) | 75 | 42
  C6D1 | 0.0594 (0.26864) | 0.0658 (0.24229)
  C7D1: number analyzed (Participants) | 69 | 22
  C7D1 | 0.0853 (0.24019) | 0.1066 (0.25848)

14. Secondary Outcome: Time to Spleen and Disease Progression Free Survival (SDPFS)
Description: Time from randomization to death due to any reason or disease progression (modified IWG-MRT 2013 including ≥ 25% increase in spleen volume by MRI/CT).
Time Frame: From randomization to the End of Survival Follow-up
Reporting Status: Not Posted, anticipated posting 2026-07

15. Secondary Outcome: Overall Survival
Description: Time from randomization to death due to any reason
Time Frame: From Randomization to the end of Survival Follow Up
Reporting Status: Not Posted, anticipated posting 2026-07

ADVERSE EVENTS:
Time Frame: Adverse Events, Serious Adverse Events and All Cause Mortality: From first dose to database lock: Approximately 3 years and 8 months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Fedratinib After Crossover: Fedratinib 400mg/day PO(4x100mg capsules) after crossing over from BAT after cycle 6
Arm/Group | Fedratinib | Best Available Therapy (BAT) | Fedratinib After Crossover
All-Cause Mortality (participants affected / at risk) | 43/134 | 7/67 | 11/46
Serious Adverse Events (participants affected / at risk) | 72/134 | 21/67 | 16/46
Other Adverse Events (participants affected / at risk) | 128/134 | 57/67 | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fedratinib (N=134) | Best Available Therapy (BAT) (N=67) | Fedratinib After Crossover (N=46)
Anaemia (Blood and lymphatic system disorders) | 9 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 4 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Adrenal haemorrhage (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Retinal oedema (Eye disorders) | 1 | 0 | 0
Uveitis (Eye disorders) | 2 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Exercise tolerance decreased (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 10 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 3 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lymph node tuberculosis (Infections and infestations) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 3 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 3
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Delirium febrile (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0
Breast fibrosis (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fedratinib (N=134) | Best Available Therapy (BAT) (N=67) | Fedratinib After Crossover (N=46)
Anaemia (Blood and lymphatic system disorders) | 55 | 24 | 19
Leukocytosis (Blood and lymphatic system disorders) | 4 | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 9 | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 48 | 12 | 13
Conjunctival haemorrhage (Eye disorders) | 2 | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 5 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 15 | 9 | 6
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5 | 1
Constipation (Gastrointestinal disorders) | 30 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 62 | 3 | 17
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 54 | 10 | 11
Vomiting (Gastrointestinal disorders) | 24 | 3 | 9
Asthenia (General disorders) | 27 | 15 | 8
Fatigue (General disorders) | 11 | 10 | 4
Oedema peripheral (General disorders) | 25 | 7 | 6
Pyrexia (General disorders) | 17 | 7 | 4
COVID-19 (Infections and infestations) | 19 | 4 | 9
Urinary tract infection (Infections and infestations) | 9 | 4 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 3
Alanine aminotransferase increased (Investigations) | 10 | 1 | 2
Blood creatinine increased (Investigations) | 17 | 1 | 4
Glomerular filtration rate decreased (Investigations) | 12 | 1 | 2
Vitamin B1 decreased (Investigations) | 17 | 2 | 4
Weight decreased (Investigations) | 9 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 17 | 9 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2 | 0
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 9 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 4
Headache (Nervous system disorders) | 15 | 4 | 2
Insomnia (Psychiatric disorders) | 7 | 4 | 2
Chronic kidney disease (Renal and urinary disorders) | 7 | 0 | 3
Renal failure (Renal and urinary disorders) | 6 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 4 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 4 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 8 | 9 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 10 | 5
Haematoma (Vascular disorders) | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03952039/Prot_SAP_000.pdf